#### ASSENT FORM FOR CHILDREN AGED 8 TO 14 YEARS

Study Title: Exposure-Response Evaluation of IV Artesunate in Children with Severe Malaria

Study short name: IV Artesunate in Children with Severe Malaria

Principal Investigator: Prof. Matthew B Laurens, MLaurens@som.umaryland.edu

Site Principal Investigator: Dr Pauline Byakika-Kibwika,

Sponsor: Division of Microbiology and Infectious Diseases, National Institute of Allergy & Infectious

Diseases, U.S. National Institutes of Health Site: Tororo District Hospital, Tororo, Uganda

Participant Study ID: M26TRH

### A. Why have we met you?

We want to tell you about something we are doing called a research study. A research study is when a group of people collect information to learn more about something. In this research study we will be learning more about a drug used to treat malaria called Artesunate. After we tell you about it, we will ask if you would like to take part in this research study or not.

# B. Why are the doctors doing this research?

This is a research study being done to learn more about the medication used to treat severe malaria (called artesunate). The team of doctors doing this research want to learn how the human body breaks down the drug artesunate when it is given into the blood vessel (intravenously) to a patient with severe malaria, how the effects of malaria in the body change when a patient receives artesunate, and the time artesunate takes to kill malaria parasites in the body. We will also learn more about how quickly artesunate helps the body functions to return to normal. Artesunate is a drug used for treatment of severe malaria in Uganda. To learn more about artesunate, we will be doing additional observations and tests that would not normally be done for patients with severe malaria at Tororo District hospital. If you do not participate, you will still be treated for malaria. If you do participate, you can change your mind at any time, and you will still be treated for malaria.

# C. What is expected of you if you are involved in this research?

1. If you accept to participate in this study, we will collect 8.25 mL (approximately 1 to 2 teaspoons) of blood at the screening visit to check if you are suitable to participate in the study. Alternatively, we may collect information from your medical records if the tests were done within the previous 24 hours. If you meet the eligibility criteria, we will collect 11.5 mL (approximately 2 to 2 ½ teaspoons) of blood at the enrolment visit and 1-3.5 mL of blood (approximately ¼ to ½ teaspoon) at other times during the study (see schedule below). If you are suitable to participate in this research, you will be seen every day for the time that you are in the hospital, up to 7 days. You will the then have up to 4 more study visits 1, 2, 4, and 26 weeks from now, which are planned to happen in the study clinic.

# 2. Screening Visit (Day -1 to 1)

After you have signed the form accepting to be in this study, you will have a physical exam, your vital signs including height and weight will be checked and you will have 8.25 mL (approximately 1 to 2 teaspoons) of blood taken to check for malaria parasites, blood counts, blood chemistry, blood artesunate level, and malaria genes that control parasite growth and development. Any medicine you are taking will be noted. A urine specimen will be collected, and you will start IV artesunate treatment for severe malaria according to the standard guidelines. Based on the results of these tests, the research staff will tell you whether you are able to enter the research or not.

### 3. Enrolment Visit (Day 1)

You will have a physical exam and vital signs will be checked, and you will have 11.5 mL (approximately 2 to 2 ½ teaspoons) of blood taken to check for malaria parasites, blood counts, blood chemistry, and blood artesunate level. A urine specimen will be collected, and you will be given your IV artesunate treatment according to standard guidelines. Enrolment is complete after these exams.

### 4. Daily Hospital Visits (Days 2 to 6)

You will have a physical exam and vital signs will be checked, and you will have 3-3.5 mL (approximately ½ teaspoon) of blood taken to check for malaria parasites, blood counts, and blood chemistry. A urine specimen will be collected. IV artesunate or oral artemisinin combination therapy will be given according to standard guidelines.

### 5. Study Visit (Day 7)

You will have a physical exam and vital signs will be checked, and you will have 3 mL (approximately ½ teaspoon) of blood taken to check for blood counts and blood chemistry. A urine specimen will be collected.

# 6. Study Visit (Day 14)

You will have a physical exam and vital signs will be checked (if needed) and we will have 3 mL (approximately ½ teaspoon) of blood taken to check for blood counts and blood chemistry.

### 7. Study Visit (Day 28)

You will have a physical exam and vital signs will be checked (if needed) and you will have 1 mL (approximately ½ teaspoon) of blood taken to check for blood counts.

# 8. Final Study Visit (Day 183)

You will have a physical exam and vital signs will be checked and you will have 1 mL (approximately ¼ teaspoon) of blood taken to check for blood counts.

In this study, we will collect blood samples from you, and we will use these samples to test how your body responds to the artesunate medicine used to treat malaria and to see how fast your body breaks down the drug, how the effects of malaria in the body change when a patient receives artesunate, and the time it takes to clear parasites from the blood. Your blood samples will be labelled only by a code and will not be labelled with your name or initials. These coded samples will be kept at a storage facility and may be shared with investigators at this institution and at other institutions. Electronic files associated with these coded samples will be password protected. Only people who are involved in this study will be allowed to see the files.

If these stored blood samples are tested in the future, the results may be shared with other researchers and the public; however, you will not be identified in these results, and none of your private information will be shared with the results. In other words, the publication will not contain any information about you that would allow someone to find out your identity. The results of any future testing will be kept private in the same way as the results of testing done for this study. Results from future research will not be reported to your doctor or be placed in your medical record. Your decision to participate can be changed at any time by telling study staff. However, we may continue to use information we got from your blood samples before you change your decision. Your decision about your blood samples will not affect your participation in other studies or your medical care.

### D. What will you gain from this research?

There may be no direct benefit of participation in the study, however the knowledge gained from this study may help the country of Uganda, Africa, and the world at large in determining the best way to give treatment for severe malaria. You will benefit by having very close monitoring of your health and treatment of severe malaria during the study period.

### E. Can this research cause harm?

You may feel pain when the sample of blood is being removed from your finger or vein, but it will subside quickly. Sometimes some questions we ask you may make you uncomfortable, but we shall make sure this does not happen many times.

If you are injured or you have questions about injuries as a result of being in the study, you can contact the doctors in the study clinic and/or Prof. Pauline Byakika-Kibwika (telephone offered at the hospital will be available in case of any such injury. Care will be provided free of charge for injuries related to study participation using study funds. In addition, we will reimburse the cost of consultation for referrals made by study physicians to other clinics and services within the hospital. The NIH will not provide any long-term medical care or any other payment for research related injuries.

## F. How long will you be in this study?

You will be in the study for 6 months (183 days), unless the doctors or your parents or guardians decide you should leave the study earlier.

### G. Do you have any questions?

You may ask questions any time either now or later. You can talk to me or somebody else. Prof Byakika and the staff are available to explain this study to you and answer your questions. If you have questions about the study, you may call Prof Byakika (Telephone ). If you have questions about your rights as a research subject, you may contact the chairman of the Infectious Diseases Institute Research Ethics Committee, Dr. David Patrick Kateete (Telephone-)

### H. Must you be in this research?

No one will force you into this research study. Do not feel ashamed to tell us. Remember you may accept now and later on refuse; however, it is your own choice if you are not interested in this study or if you change your mind later. You will receive medical care if you are sick whether or not you are in the study. Let us know whether you have accepted or not.

The research staff will give you a copy of this agreement

#### I. Will I be paid for taking part in this study?

You will not be paid to participate in the study. We will provide a refund of 20,000 UGX for transport costs on scheduled study visits.

# Assent to Join the Research

The study has been explained to me in a language I can understand. I have had the opportunity to ask questions about it and my questions have been answered to my satisfaction. I assent voluntarily to be in the study.

Put your initials/thumbprint in the boxes at the end of each statement

| 1 | I have read/been read the assent form. I have had the opportunity to ask questions about this study and I am satisfied with the answers that I have been given. | |
|---|---|---|
| 2 | I agree to be asked questions about my health | |
| 3 | I understand some testing of samples will be tested overseas and I agree that specimens be sent for this. | |
| 4 | I understand that my participation is voluntary and will have no effect on my medical treatment. I understand that I can withdraw from the study at any time. | |
| 1 | Name of participant | |
| Signature or thumbprint of participant | | |
| I | Date of Signature Day/month/year | |
| I | filliterate | Thumbprint |
| A literate witness must sign (if possible, this person should be selected by the participant and should have no connection to the research team and should not be a relative to the participant). Participants who are illiterate should include their thumbprint as well. | | |
| 5 | Statement by the witness | |
| | have witnessed the accurate reading of the assent form to the potential participant, a apportunity to ask questions. I confirm that the individual has given assent freely. | and the individual has had the |
| 1 | Name of witness | |
| 5 | Signature of witness | |
| Ι | Date of Signature Dav/Month/Year | |

### Statement by the researcher taking assent:

The informed assent document has been read by/been read aloud to the potential study participant. To the best of my ability, I have ensured that the participant understands

- 1. The reasons for the study/studies
- 2. The sampling and follow-up arrangements for participation
- 3. Plans for protection of confidential data and dissemination of results

I confirm that the participant was given an opportunity to ask questions about the study, and all questions have been answered correctly and to the best of my ability. I confirm that assent has been given freely and voluntarily.

| Name of Researcher/Person taking the Assent | t |
|----------------------------------------------|------|
| Signature of Researcher/Person taking the As | sent |
| Date: | |
| Day/Month/Year | |